CLINICAL TRIAL: NCT03666273
Title: An Open-label, Phase 1, First-in-human, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Maximum Tolerated or Administered Dose, Pharmacokinetics, Pharmacodynamics and Tumor Response Profile of the ILDR2 Function-blocking Antibody BAY1905254 in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Study of BAY1905254 - An Early Clinical Research Study to Evaluate a New Drug Called Bapotulimab (BAY1905254) in the Expansion Cohort in Combination With Pembrolizumab in Head and Neck Cancer That Has Returned or is Discovered to be Metastatic and is Expressing PDL1.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18789; MK-3475-920 (Other: Merck Sharp & Dohme LLC); KEYNOTE-920 (Other: Merck Sharp & Dohme LLC); 2018-000990-63 (EudraCT Number)
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor; Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Head and Neck Cancer; Immunotherapy; PD1, PDL1, ILDR2; Bapotulimab; Pembrolizumab; Immune checkpoint inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation_Monotherapy (Experimental): Patients with solid tumor types considered immunosensitive
  Interventions: Drug: Bapotulimab (BAY1905254)
- Dose escalation_Combination therapy (Experimental): Patients with solid tumor types considered immunosensitive
  Interventions: Drug: Bapotulimab (BAY1905254) + Pembrolizumab (KEYTRUDA®)
- Expansion HNSCC_Combination therapy (Experimental): Patients with head and neck squamous cell carcinoma (HNSCC)
  Interventions: Drug: Bapotulimab (BAY1905254) + Pembrolizumab (KEYTRUDA®)

INTERVENTIONS:
Drug: Bapotulimab (BAY1905254) — Intravenous administration of escalating doses of Bapotulimab
  Arms: Dose escalation_Monotherapy
Drug: Bapotulimab (BAY1905254) + Pembrolizumab (KEYTRUDA®) — Intravenous administration of Bapotulimab of fixed dose (expansion), and of a fixed dose of pembrolizumab
  Arms: Dose escalation_Combination therapy; Expansion HNSCC_Combination therapy

SUMMARY:
This study is being done to learn more about a new drug called Bapotulimab given in combination with Pembrolizumab. The purpose of this study is to learn if this new combination of drugs is safe for the participants, how it affects the body and to try to find the best dose of the new drug to give to participants and to obtain a preliminary assessment of the tumor response efficacy in the recurrent or metastatic Head and Neck Cancer.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients aged ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Patients must have measurable disease (at least one unidimensional measurable lesion by Computed tomography [CT] or Magnetic resonance imaging [MRI]) per Response evaluation criteria in solid tumors (RECIST) 1.1, and following histologically confirmed, advanced or metastatic solid tumors:

  * Dose escalation: All solid tumor types with a likelihood of sensitivity to immunotherapy, as judged by the investigator.
  * Expansion of Bapotulimab in combination with pembrolizumab in Head and neck squamous cell carcinoma (HNSCC): recurrent or metastatic head and neck squamous cell carcinoma IO-naïve PDL1+/ CPS≥1(PD-L1: Programmed death ligand 1; CPS: Combined positive score).
* Provision of archival tumor tissue at screening is mandatory for all patients in dose escalation.
* For dose escalation, patients: must have received standard therapy or have no standard therapy available or patients have actively refused any treatment which would be regarded standard. Or in the opinion of investigator have been considered ineligible for a particular form of standard therapy on medical grounds.
* Adequate bone marrow, liver and renal function.
* Adequate cardiac function, measured by echocardiography.

Main Exclusion Criteria:

* History of severe immune related adverse effects from prior immunotherapy (CTCAE v.5.0 Grade 4; CTCAE v.5.0 Grade 3 requiring treatment > 4 weeks), except hypothyroidism clinically stable on hormone replacement treatment and controlled type 1 diabetes.
* Severe (CTCAE v.5.0 Grade ≥ 3) infections within 4 weeks before the first study drug administration, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia. Clinically active infections (CTCAE v.5.0 > Grade 1) within 2 weeks before the first study drug administration.
* Previous or active myocarditis/myositis in history (independent of cause)
* Active or history of autoimmune disease.
* Known human immunodeficiency virus (HIV) infection.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Treatment with systemic immunosuppressant medications within 2 weeks before the first study drug administration.
* Ongoing or previous anti-cancer treatment or any immunostimulatory treatment including but not limited to interferons (IFNs), interleukin (IL)-2 and agonists for members of the tumor necrosis factor (TNF) receptor superfamily (e.g. 4-1BB) within 4 weeks before the first study drug administration.
* For dose expansion cohort of Bapotulimab in combination with pembrolizumab in HNSCC: has progressive disease (PD) within six (6) months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs (TEAEs) including treatment-emergent serious adverse events (TESAEs), adverse events of special interest (AESIs), and dose-limiting toxicities (DLTs) | Up to 58 months
Severity of treatment-emergent AEs (TEAEs) including treatment-emergent serious adverse events (TESAEs), adverse events of special interest (AESIs), and dose-limiting toxicities (DLTs) | Up to 58 months
Cmax of Bapotulimab after first dose administration (Cycle 1) for cohorts receiving doses ≥ 20 mg | Up to 504 hours after drug in Cycle 1
  Maximum plasma concentration after single dose
AUC of Bapotulimab after first dose administration (Cycle 1) for cohorts receiving doses ≥ 20 mg | Up to 504 hours after drug in Cycle 1
  Area under the plasma concentration curve after single dose
Maximum tolerated dose (MTD) of Bapotulimab | Up to 58 months

SECONDARY OUTCOMES:
Recommended dose of Bapotulimab for Phase 2 | Up to 58 months
Cmax,md after multiple dosing (Cycle 3) for cohorts receiving doses ≥ 20 mg | Up to 504 hours after drug in Cycle 3
  Maximum plasma concentration after multiple doses
AUC after multiple dosing (Cycle 3) for cohorts receiving doses ≥ 20 mg | Up to 504 hours after drug in Cycle 3
  Area under the plasma concentration curve after multiple doses
Incidence of positive anti-drug antibody titer for Bapotulimab | Up to 58 months
Best overall response rate | Up to 58 months
  Determined by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- United States (8):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Chicago Hospitals, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics | START San Antonio, San Antonio, Texas